CLINICAL TRIAL: NCT00588757
Title: Prospective Comparison Between OptEase and Gunter-Tulip
Brief Title: Comparison Between Two Optional IVC Filters Regardind Ease of Use,Complications and Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Uri Rimon, Sehba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-07-4741-UR-CTIL
Record Dates: First submitted 2007-12-25; First posted 2008-01-09 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: Trauma; Deep Vein Thrombosis
Keywords: IVC filters; Trauma; Dwell time
MeSH Terms: conditions — Wounds and Injuries; Venous Thrombosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Optease filter
  Interventions: Device: Optease IVC filters
- 2 (Active Comparator): Tulip filter
  Interventions: Device: Gunter-Tulip IVC filters

INTERVENTIONS:
Device: Optease IVC filters — IVC filters will be implemented and evaluated for retrieval after 2-3 weeks.
  Arms: 1
Device: Gunter-Tulip IVC filters — IVC filters will be implemented and evaluated for retrieval after 2-3 weeks.
  Arms: 2

SUMMARY:
OptEase filters are easier to retrieve but the dwell time is shorter than the Gunter filters. There are more thrombi on the OptEase than on the Gunter at the time of retrieval. OptEase filter has a better infitration capabillity due to its diamond shape. OptEase filters will hjave more IVC occlusions as a complication.

DETAILED DESCRIPTION:
We will isert the two filters blindly. We will follow the patients clinically and if needed we will add imaging exams. We will try to retrieve most filters.

ELIGIBILITY:
Inclusion Criteria:

* All patients referred for filter insertion

Exclusion Criteria:

* Young age (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
comparing the two filters | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Uri Rimon, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel